CLINICAL TRIAL: NCT01126229
Title: A Pilot Study of Resveratrol Supplementation for Memory and Physical Performance
Brief Title: Resveratrol for Improved Performance in the Elderly
Acronym: RIPE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 238-2009
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Memory
Keywords: Resveratrol; Grape; Aging; functional MRI (fMRI); Anti-Aging therapeutic; Oxidative Stress; Functional Performance
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Dietary Supplement: placebo
  Interventions: Dietary Supplement: Placebo
- 300 mg/d Resveratrol (Experimental): Dietary Supplement: 300 mg/d Resveratrol
  Interventions: Drug: Low dose Resveratrol
- 1000 mg/d Resveratrol (Experimental): Dietary Supplement: 1000 mg/d Resveratrol
  Interventions: Drug: High dose Resveratrol

INTERVENTIONS:
Dietary Supplement: Placebo — 2 capsules of placebo daily for 12 weeks
  Arms: Placebo
Drug: Low dose Resveratrol — 2 capsules daily for 12 weeks containing 300 mg/d (combined) of resveratrol active ingredient
  Other Names: ReserveAge
  Arms: 300 mg/d Resveratrol
Drug: High dose Resveratrol — 2 capsules daily for 12 weeks containing 1000 mg/d (combined) of resveratrol active ingredient
  Other Names: ReserveAge
  Arms: 1000 mg/d Resveratrol

SUMMARY:
The investigators aim to conduct a randomized placebo controlled pilot study to determine whether resveratrol, a dietary ingredient, supplementation is safe and improves memory and physical performance in older adults. Loss in memory and physical performance is a frequent complaint in older adults and a growing public health issue. Additionally, later adulthood is associated with a normative decline in both working and primary memory as well as domains including attention, speed of processing and executive function. Resveratrol is safely tolerated in pre-clinical models and in dose-escalation human studies. It also has demonstrated beneficial effects on memory and performance in pre-clinical models. Therefore, this study will take the next step in understanding the longer-term safety (3 months) and efficacy of resveratrol supplementation on age-related health conditions.

DETAILED DESCRIPTION:
Enrolled participants will complete psychological questionnaires and a multi-measure cognitive test battery, physical function, as well as provide blood samples, to determine blood chemistry. These will include complete blood count and complete metabolic count [(Na, K, Cl, CO2, BUN, Creatinine, Glucose, Total Protein, Albumin, Calcium, Phosphorous, Aspartate Aminotransferase (AST), Alkaline Phos, Total Bilirubin, and Alanine Amino Transferase (ALT)] and any others deemed necessary by the study physician. They will return to the laboratory to perform a muscular endurance test and MRI evaluation at the Brain Institute. Eligible participants will be randomly assigned with equal probability to either receive resveratrol (300 mg/d or 1000 mg/d) or placebo for twelve weeks. Immediately following completion of the MRI, participants will be given a month's supply of resveratrol or placebo. All participants will be closely monitored for safety and toxicity during the first 10 days (range 8-12 days are acceptable) of the trial. During this initial evaluation period, blood chemistries (complete metabolic profiles) will be evaluated every 3 (range 1-2 days are acceptable) days. Following one month, participants will be asked to return to clinic. At their monthly visits, memory tests, blood samples will be collected to monitor cognitive adaptations and ensure that no adverse changes have occurred. Participants' compliance with the supplementation regimen will also be checked through pill counts, and participants will be given a month's supply of product at each of their monthly visits. After 12 weeks of taking either resveratrol or a placebo on a daily basis, participants will complete a final test battery, an MRI scan, a blood draw collection. A follow-up evaluation will be provided at 10 and 30 days following completion of the final post-treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65-100 years
* Body mass index > = 25 and < = 35
* Willing and able to participate in all aspects of the study
* Willing to be randomized to either treatment group
* Sedentary to moderately active lifestyle (<120 min aerobic activity/week)
* Report of ability to walk one mile
* MMSE > 24
* Non-smoking
* Telephone Interview for cognitive status (TICS)

Exclusion Criteria:

* Active treatment for cancer, stroke (< 6 mo), peripheral vascular disease, coronary artery disease (myocardial infarction <6 mo), state III, IV Congestive Heart Failure, valvular heart disease, major psychiatric disease, severe anemia, liver or renal disease, diabetes, severe osteoarthritis, blindness or deafness, fracture in upper or lower extremity within the last 6 months, upper or lower extremity amputation, anticoagulant therapy (aspirin use is permitted), parkinsons disease
* Failure to give consent
* Anabolic medications (growth hormone or testosterone)
* High amounts of physical activity (i.e. running, bicycling etc) > 120 min/week.
* Dementing illness
* Excessive alcohol use (>2 drinks per day)
* Resting heart rate > 120 bpm
* Systolic blood pressure > 180 mmHg
* Diastolic blood pressure > 100 mmHg
* Dietary supplementation of grape seed extract or ginko biloba
* History of significant head injury
* Vision or hearing impairment
* Anticholinesterase inhibitor (such as Aricept)
* Contraindications to MRI (e.g. cardiac pacemaker, implanted cardiac defibrillator, aneurysm clip, claustrophobia, etc.)
* Consumption of red wine/dealcoholized red wine/red or purple grape juice more than once weekly; consumption of any dietary supplements containing resveratrol, quercetin, or P. cuspidatum in the previous 90 days;
* Subject is participating in another clinical trial or has received an investigational product within 30 days prior to screening/enrollment
* Current Use of Antidepressant Medications
* CES-D Score > 20

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety Outcomes | 24 months
  CBC, Complete Metabolic Panel, Toxicity according to NCI criteria

SECONDARY OUTCOMES:
Cognitive Outcomes | 24 months
  Executive function measured by N-back and Controlled Oral Word Association test, Processing Speed measuring by Trails A & B, Memory Function measured by word recall.
Physical Outcomes | 24 months
  Physical function measured by performance on the 400 meter walk test, physical activity levels as measured by accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Manini, PhD, Principal Investigator — University of Florida, Aging and Geriatric Research; Stephen M Manini, PhD, Principal Investigator — University of Florida, Aging and Geriatric Research
Locations (1):
- University of Florida, Aging and Geriatric Research, Gainesville, Florida, United States

REFERENCES:
- [Derived] Anton SD, Embry C, Marsiske M, Lu X, Doss H, Leeuwenburgh C, Manini TM. Safety and metabolic outcomes of resveratrol supplementation in older adults: results of a twelve-week, placebo-controlled pilot study. Exp Gerontol. 2014 Sep;57:181-7. doi: 10.1016/j.exger.2014.05.015. Epub 2014 May 24. PMID 24866496